CLINICAL TRIAL: NCT01796236
Title: Clinical and Health Economic Evaluation of a New Baha® Abutment, With a Minimally Invasive Surgical Technique. An International Multicentre, Open, Randomised, Comparative, Parallel Group, Investigation. 1y Investigation, 2y Follow-up
Brief Title: Clinical and Health Economic Evaluation With a New Baha® Abutment Combined With a Minimally Invasive Surgical Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear Bone Anchored Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBAS5439
Record Dates: First submitted 2013-01-16; First posted 2013-02-21 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Deafness; Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural
Keywords: Bone anchored hearing aid; Bone anchored implant; Abbreviated Profile of Hearing Aid Benefit (APHAB); Health Utility Index (HUI); Holgers Index; Implant stability
MeSH Terms: conditions — Deafness; Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimally invasive surgery and BA400 (Active Comparator): This arm involves no soft tissue reduction around the BA400 implant.
  Interventions: Device: Minimally invasive surgery and BA400
- Traditional surgery and BA300 (Active Comparator): This arm involves traditional soft tissue reduction around the BA300 implant
  Interventions: Device: Traditional surgery and BA300

INTERVENTIONS:
Device: Minimally invasive surgery and BA400 — The Cochlear Baha BA400 Abutment has been designed with a concave shape at the lower aspect of the abutment. The abutment is made of commercially pure titanium and is coated with a hydroxyapatite layer on the entire soft tissue-contacting surface of the abutment up to 3 mm below the top surface (2 mm below the top surface on 6 mm abutments).
  Arms: Minimally invasive surgery and BA400
Device: Traditional surgery and BA300 — The BA300 abutment is made of commercially pure titanium and is available in two different lengths (6 mm and 9 mm).
  Arms: Traditional surgery and BA300

SUMMARY:
To demonstrate that the minimally invasive surgical procedure in combination with the use of the Cochlear Baha BA400 abutment is associated with a reduction of inflammation/infection, overgrowth, pain and numbness at the site of implantation compared to the traditional surgical procedure in combination with the use of the standard Baha abutment (Cochlear Baha BA300 Abutment).

To demonstrate that the minimally invasive surgical procedure in combination with the use of the Cochlear Baha BA400 abutment is associated with a reduction in direct medical costs, due to shorter surgical procedures, faster wound healing and less complications compared to the traditional surgical procedure in combination with the use of the standard Baha abutment (Cochlear Baha BA300 Abutment).

DETAILED DESCRIPTION:
Despite extensive soft tissue reduction, the most common complications associated with Baha implants are related to adverse skin reactions around the abutment. The reduction of the skin also adds complexity to the surgical procedure that is otherwise a routine type of skin incision. A less invasive surgical technique avoiding reducing the thickness of the skin would render a simpler and shorter procedure and would be aesthetically appealing to the patients, as permanent hair removal in the area around the abutment would not be required. Faster healing and less numbness (sensory loss/ paraesthesia) at the implant site may also be expected if the soft tissue thickness is left intact.

The Cochlea Baha BA300 Abutment together with a surgical procedure that includes soft tissue reduction was CE marked in April 2010. The test abutment, Cochlear Baha BA400, together with a surgical procedure that does not require soft tissue reduction was CE marked in June 2012.

The rationale behind this investigation was to make a 'head-to-head' comparison between the BA300 and BA400 Abutment and the associated surgical techniques in order to collect information regarding complications (inflammation/infection, numbness and pain), aesthetic outcome and utilisation of direct medical cost associated with surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for the Baha system
* Signed informed consent

Exclusion Criteria:

* Patient scheduled for simultaneously bilateral implant surgery
* Uncontrolled diabetes as judged by the investigator
* Condition that could jeopardize osseointegration and/or wound healing, e.g. osteoporosis, psoriasis and use of corticosteroids
* Unable to follow the cleaning instruction
* Unable to follow investigational procedures, e.g. to complete quality of life scales
* Participation in another investigation with pharmaceuticals and/or device
* Condition that may have an impact on the outcome of the investigation as judged by the investigator
* Suitable implant position for the 4 mm implant not found during surgery due to insufficient bone quality and/or bone thickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stokroos, Professor, Principal Investigator — NT department, Oxford Building , Peter Debyelaan 25, 6202 AZ Maastricht, The Netherlands
Locations (7):
- Service ORL, Toulouse, France
- Netherlands (4):
  - KNO arts, Amphia Ziekenhuis, Breda
  - Deventer Ziekenhuis, Deventer
  - Dept. ENT/KNO, Eindhoven
  - NT department, Maastricht
- Otorhinolaryngology, Hospital Clinico Universitario De Valencia, Valencia, Spain
- ENT Clinic, Gothenburg, Sweden

REFERENCES:
- [Derived] van Hoof M, Wigren S, Ivarsson Blechert J, Molin M, Andersson H, Mateijsen DJM, Bom SJH, Calmels MN, van der Rijt AJM, Flynn MC, van Tongeren J, Hof JR, Brunings JW, Anteunis LJC, Marco Algarra J, Stokroos RJ, Joore MA. A Multinational Cost-Consequence Analysis of a Bone Conduction Hearing Implant System-A Randomized Trial of a Conventional vs. a Less Invasive Treatment With New Abutment Technology. Front Neurol. 2020 Mar 13;11:106. doi: 10.3389/fneur.2020.00106. eCollection 2020. PMID 32231633

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 106 subjects signed informed consent. Before surgery one subject cancelled surgery, one subject withdraw consent and one subject got the wrong allocation due to logistic problems. This resulted in that 103 subjects received the allocated intervention (51 test and 52 control).
Groups:
- Minimally Invasive Surgery and BA400: This arm involves no soft tissue reduction around the BA400 implant.
  Minimally invasive surgery and BA400: The Cochlear Baha BA400 Abutment has been designed with a concave shape at the lower aspect of the abutment. The abutment is made of commercially pure titanium and is coated with a hydroxyapatite layer on the entire soft tissue-contacting surface of the abutment up to 3 mm below the top surface (2 mm below the top surface on 6 mm abutments). The abutment is available in four different lengths (6, 8, 10 and 12 mm)
Period: Overall Study
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Started | 51 | 52
Completed | 49 | 50
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300 | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (10.9) | 51.5 (16.6) | 52.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 26 | 25 | 51
Region of Enrollment [Number; unit: participants]
  Netherlands | 26 | 29 | 55
  Sweden | 5 | 4 | 9
  France | 5 | 5 | 10
  Spain | 15 | 14 | 29
Use of nicotine [Number; unit: participants]
  No | 37 | 38 | 75
  Yes | 14 | 13 | 27
  Unknown | 0 | 1 | 1
Type of hearing loss [Number; unit: participants]
  Conductive | 5 | 10 | 15
  Mixed | 31 | 35 | 66
  Single-Sided Sensorineural | 15 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Adverse Events as a Measure of Safety and Tolerability
Description: Combined endpoint of infection/inflammation, overgrowth, pain and numbness will be evaluated, as the sum of the following four events:
  1. Holgers Index >=2 any time between 3 weeks to 1 year
  2. Any overgrowth any time between 3 weeks to 1 year
  3. Pain (scar/neuropathic) according to POSAS >=3 any time between 3 weeks to 1 year
  4. Any numbness any time between 3 weeks to 1 year Each medical event is counted only once per subject resulting in a score of 0 to 4 for every subject.
Time Frame: 12 months
Population: The Intent-to-Treat population (ITT) consisted of all randomised patients with at least one follow-up measurement from visit 3 Day 10 and onward.
Measure: Number; unit: participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
participants
  Combined endpoint score = 0 | 15 | 7
  Combined endpoint score = 1 | 14 | 13
  Combined endpoint score = 2 | 14 | 24
  Combined endpoint score = 3 | 7 | 8
  Combined endpoint score = 4 | 1 | 0
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Test type: Superiority or Other; p = 0.12, Mantel Haenszel

2. Primary Outcome: Number of Participants With Local Adverse Events as a Measure of Safety and Tolerability
Description: as for outcome 1
Time Frame: 36 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
participants
  Combined endpoint score = 0 | 12 | 5
  Combined endpoint score = 1 | 12 | 15
  Combined endpoint score = 2 | 16 | 23
  Combined endpoint score = 3 | 9 | 8
  Combined endpoint score = 4 | 2 | 1
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Combined Endpoint is calculated as the sum of the following four events from 3 weeks to 3 years: Holgers Index >=2. Any Overgrowth >=2. Pain (scar/neuropathic) >=3. Any numbness >=2. Each event is counted only once; Test type: Superiority or Other; p = 0.45, Mantel Haenszel

3. Secondary Outcome: Surgery Time
Description: Surgery time (minutes) was recorded
Time Frame: Day 0
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
minutes | 15.3 (6.2) | 24.7 (8.6)
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Test type: Superiority or Other; p < 0.0001, Mann-Whitney U test

4. Secondary Outcome: Wound Healing
Description: A surgeon or a surgical nurse determined if the wound was healed or not healed.
Time Frame: Day 10, Weeks 3, 6, 12 and 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
participants
  Day 10, Wound not healed | 4 | 14
  Day 10, Wound healed | 47 | 38
  Week 3, Wound not healed: number analyzed (Participants) | 50 | 52
  Week 3, Wound not healed | 4 | 8
  Week 3, Wound healed: number analyzed (Participants) | 50 | 52
  Week 3, Wound healed | 46 | 44
  Week 6, Wound not healed: number analyzed (Participants) | 50 | 51
  Week 6, Wound not healed | 3 | 3
  Week 6, Wound healed: number analyzed (Participants) | 50 | 51
  Week 6, Wound healed | 47 | 48
  Week 12, Wound not healed: number analyzed (Participants) | 47 | 50
  Week 12, Wound not healed | 1 | 0
  Week 12, Wound healed: number analyzed (Participants) | 47 | 50
  Week 12, Wound healed | 46 | 50
  Week 24, Wound not healed: number analyzed (Participants) | 47 | 46
  Week 24, Wound not healed | 0 | 0
  Week 24, Wound healed: number analyzed (Participants) | 47 | 46
  Week 24, Wound healed | 47 | 46
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Day 10; Test type: Superiority or Other; p = 0.020, Fisher Exact
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 3; Test type: Superiority or Other; p = 0.4, Fisher Exact
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 6; Test type: Superiority or Other; p = 1.00, Fisher Exact
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12; Test type: Superiority or Other; p = 0.97, Fisher Exact
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24; Test type: Superiority or Other; p = 1.00, Fisher Exact

5. Secondary Outcome: Inflammation - Max of Holgers Index
Description: Max of Holgers index from day 10 to month 12, and to month 36 was recorded, using the Holgers scale from 0 - 4, where 0 = no inflammation and 4 = removal of abutment/implant necessary due to infection.
  0. No irritation
  1. Slight redness. Local temporary treatment, if needed
  2. Red and slightly moist tissue. No granulation formation, local treatment and extra controls as indicated*
  3. Reddish and moist; sometimes granulations tissue, revision surgery is indicated* R. Removal of the abutment / implant necessary due to infection* R Removal of implant for reasons not related to skin problems*
Time Frame: From Day 10 to 12 Months, and to 36 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
Participants
  Max of Holgers 12 Months: Max of Holgers index = 0 | 10 | 8
  Max of Holgers 12 Months: Max of Holgers index = 1 | 26 | 32
  Max of Holgers 12 Months: Max of Holgers index = 2 | 7 | 10
  Max of Holgers 12 Months: Max of Holgers index = 3 | 8 | 2
  Max of Holgers 12 Months: Max of Holgers index = 4 | 0 | 0
  Max of Holgers 36 Months: Max of Holgers index = 0 | 9 | 8
  Max of Holgers 36 Months: Max of Holgers index = 1 | 23 | 31
  Max of Holgers 36 Months: Max of Holgers index = 2 | 7 | 9
  Max of Holgers 36 Months: Max of Holgers index = 3 | 11 | 4
  Max of Holgers 36 Months: Max of Holgers index = 4 | 1 | 0
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Maximum of Holgers at 12 Months; Test type: Superiority or Other; p = 0.40, Mantel Haenszel
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Maximum of Holgers at 36 Months; Test type: Superiority or Other; p = 0.14, Mantel Haenszel

6. Secondary Outcome: Inflammation - Holgers Index by Visit
Description: Infection and inflammation were evaluated by the holgers index at visits 3-10 (Day 10, Weeks 3, 6, 12, 24, months 12, 24 and 36) and the following scale was used:
  0. No irritation. Epidermal debris removed, if present
  1. Slight redness. Local temporary treatment, if needed
  2. Red and slightly moist tissue. No granulation formation, local treatment and extra controls as indicated*
  3. Reddish and moist; sometimes granulations tissue, revision surgery is indicated*
  4. Removal of the abutment / implant necessary due to infection* R. Removal of implant for reasons not related to skin problems*
Time Frame: Day 10, Weeks 3, 6, 12, 24, months 12, 24 and 36
Population: The Intent-to-Treat population (ITT) consisted of all randomised patients with at least one follow-up measurement from visit 3 Day 10 through to month 36.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
Participants
  Day 10: Holgers 0 | 32 | 35
  Day 10: Holgers 1 | 15 | 15
  Day 10: Holgers 2 | 2 | 2
  Day 10: Holgers 3 | 2 | 0
  Day 10: Holgers 4/ Removal | 0 | 0
  Week 3: number analyzed (Participants) | 50 | 52
  Week 3: Holgers 0 | 27 | 33
  Week 3: Holgers 1 | 17 | 16
  Week 3: Holgers 2 | 2 | 2
  Week 3: Holgers 3 | 4 | 1
  Week 3: Holgers 4/ Removal | 0 | 0
  Week 6: number analyzed (Participants) | 50 | 51
  Week 6: Holgers 0 | 32 | 29
  Week 6: Holgers 1 | 17 | 18
  Week 6: Holgers 2 | 0 | 3
  Week 6: Holgers 3 | 0 | 1
  Week 6: Holgers 4/ Removal | 1 | 0
  Week 12: number analyzed (Participants) | 47 | 50
  Week 12: Holgers 0 | 33 | 36
  Week 12: Holgers 1 | 11 | 12
  Week 12: Holgers 2 | 3 | 2
  Week 12: Holgers 3 | 0 | 0
  Week 12: Holgers 4/ Removal | 0 | 0
  Week 24: number analyzed (Participants) | 47 | 46
  Week 24: Holgers 0 | 32 | 27
  Week 24: Holgers 1 | 13 | 17
  Week 24: Holgers 2 | 2 | 2
  Week 24: Holgers 3 | 0 | 0
  Week 24: Holgers 4/ Removal | 0 | 0
  Month 12: number analyzed (Participants) | 48 | 48
  Month 12: Holgers 0 | 41 | 39
  Month 12: Holgers 1 | 4 | 9
  Month 12: Holgers 2 | 1 | 0
  Month 12: Holgers 3 | 2 | 0
  Month 12: Holgers 4/ Removal | 0 | 0
  Month 24: number analyzed (Participants) | 46 | 46
  Month 24: Holgers 0 | 37 | 40
  Month 24: Holgers 1 | 8 | 6
  Month 24: Holgers 2 | 0 | 0
  Month 24: Holgers 3 | 0 | 0
  Month 24: Holgers 4/ Removal | 1 | 0
  Month 36: number analyzed (Participants) | 45 | 41
  Month 36: Holgers 0 | 38 | 37
  Month 36: Holgers 1 | 5 | 2
  Month 36: Holgers 2 | 0 | 0
  Month 36: Holgers 3 | 2 | 2
  Month 36: Holgers 4/ Removal | 0 | 0
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Holgers Index Day 10; Test type: Superiority or Other; p = 0.38, Mantel Haenszel
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Holgers Index Week 3; Test type: Superiority or Other; p = 0.17, Mantel Haenszel
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Holgers Index Week 6; Test type: Superiority or Other; p = 0.37, Mantel Haenszel
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Holgers Index Week 12; Test type: Superiority or Other; p = 0.73, Mantel Haenszel
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Holgers Index Week 24; Test type: Superiority or Other; p = 0.47, Mantel Haenszel
Statistical Analysis 6: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Holgers Index Month 12; Test type: Superiority or Other; p = 0.73, Mantel Haenszel
Statistical Analysis 7: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Holgers Index Month 24; Test type: Superiority or Other; p = 0.37, Mantel Haenszel
Statistical Analysis 8: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Holgers Index Month 36; Test type: Superiority or Other; p = 0.75, Mantel Haenszel

7. Secondary Outcome: Max Numbness
Description: Subjects were asked if they experience any numbness around the abutment at each visit. The maximum numbness each subject experienced is summarized in this analysis. The following scale will be used:
  1. No numbness
  2. Numbness within 2 cm from the abutment
  3. Numbness within and beyond 2 cm from the abutment
Time Frame: 12 & 36 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
Participants
  Max Numbness 12 months: No numbness | 27 | 9
  Max Numbness 12 months: Numbness within 2 cm from the abutment | 17 | 12
  Max Numbness 12 months: Numbness within and beyond 2 cm from the abutment | 7 | 31
  Max Numbness 36 months: No numbness | 27 | 9
  Max Numbness 36 months: Numbness within 2 cm from the abutment | 16 | 12
  Max Numbness 36 months: Numbness within and beyond 2 cm from the abutment | 8 | 31
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; maximum numbness at 12 months; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; maximum numbness at 36 months; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel

8. Secondary Outcome: Pain in the Scar and Neuropathic Pain
Description: The subject rated the following questions 'has the scar been painful the past few weeks' and 'have you had any neuropathic pain during the past weeks' on the 1-10 scale were 1 = no, not at all and 10 = yes, very much.
Time Frame: Day 10, Weeks 3, 6, 12, 24, Months 12 and 36
Population: The Intent-to-Treat population (ITT) consisted of all randomised patients with at least one follow-up measurement from visit 3 Day 10 and through until visit 10 Month 36.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
units on a scale
  Day 10, Neuropathic pain | 1.45 (1.47) | 1.65 (1.75)
  Day 10, Scar pain | 1.90 (1.94) | 2.08 (1.64)
  Week 3, Neuropathic pain: number analyzed (Participants) | 50 | 52
  Week 3, Neuropathic pain | 1.38 (1.26) | 1.75 (1.43)
  Week 3, Scar pain: number analyzed (Participants) | 50 | 52
  Week 3, Scar pain | 1.78 (1.52) | 1.71 (1.24)
  Week 6, Neuropathic pain: number analyzed (Participants) | 50 | 51
  Week 6, Neuropathic pain | 1.18 (0.72) | 1.45 (1.19)
  Week 6, Scar pain: number analyzed (Participants) | 50 | 51
  Week 6, Scar pain | 1.58 (1.14) | 1.80 (1.34)
  Week 12, Neuropathic pain: number analyzed (Participants) | 47 | 50
  Week 12, Neuropathic pain | 1.06 (0.25) | 1.70 (1.53)
  Week 12, Scar pain: number analyzed (Participants) | 47 | 50
  Week 12, Scar pain | 2.00 (1.41) | 2.06 (1.63)
  Week 24, Neuropathic pain: number analyzed (Participants) | 47 | 46
  Week 24, Neuropathic pain | 1.19 (0.82) | 1.41 (1.48)
  Week 24, Scar pain: number analyzed (Participants) | 47 | 46
  Week 24, Scar pain | 1.70 (1.25) | 2.02 (1.72)
  Month 12, Neuropathic pain: number analyzed (Participants) | 48 | 48
  Month 12, Neuropathic pain | 1.26 (1.05) | 1.77 (1.97)
  Month 12, Scar pain: number analyzed (Participants) | 48 | 48
  Month 12, Scar pain | 2.04 (2.01) | 2.02 (1.93)
  Month 36, Neuropathic pain: number analyzed (Participants) | 45 | 41
  Month 36, Neuropathic pain | 1.11 (0.53) | 1.39 (1.14)
  Month 36, Scar pain: number analyzed (Participants) | 45 | 41
  Month 36, Scar pain | 1.98 (1.88) | 2.05 (1.83)
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Day 10, Neuropathic pain; Test type: Superiority or Other; p = 0.74, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Day 10, Scar pain; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 3, Neuropathic pain; Test type: Superiority or Other; p = 0.030, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 3, Scar pain; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 6, Neuropathic pain; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 6, Scar pain; Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12, Neuropathic pain; Test type: Superiority or Other; p = 0.015, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12, Scar pain; Test type: Superiority or Other; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24, Neuropathic pain; Test type: Superiority or Other; p = 0.44, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24, Scar pain; Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12, Neuropathic pain; Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12, Scar pain; Test type: Superiority or Other; p = 0.97, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36, Neuropathic pain; Test type: Superiority or Other; p = 0.19, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36, Scar pain; Test type: Superiority or Other; p = 0.77, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Pain - Maximum of Neuropathic and Scar Pain
Description: The maximum neuropathic pain and the maximum scar pain experienced at any time throughout the study up until and including 12 months.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
Participants
  Neuropathic Pain: 1 - No Pain | 34 | 27
  Neuropathic Pain: 2-3 - Mild Pain | 7 | 8
  Neuropathic Pain: 4-6 - Moderate Pain | 7 | 9
  Neuropathic Pain: 7-10 - Severe Pain | 3 | 8
  Scar Pain: 1 - No Pain | 10 | 10
  Scar Pain: 2-3 - Mild Pain | 22 | 15
  Scar Pain: 4-6 - Moderate Pain | 12 | 21
  Scar Pain: 7-10 - Severe Pain | 7 | 6
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Neuropathic Categorical Max Pain; Test type: Superiority or Other; p = 0.076, Mantel Haenszel
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Scar Categorical Max Pain; Test type: Superiority or Other; p = 0.49, Mantel Haenszel

10. Secondary Outcome: Pain - Maximum of Neuropathic and Scar Pain
Description: The maximum neuropathic pain and the maximum scar pain experienced at any time throughout the study up until and including 36 months.
Time Frame: 36 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
Participants
  Neuropathic Pain: 1 - No Pain | 34 | 27
  Neuropathic Pain: 2-3 - Mild Pain | 7 | 8
  Neuropathic Pain: 4-6 - Moderate Pain | 7 | 9
  Neuropathic Pain: 7-10 - Severe Pain | 3 | 8
  Scar Pain: 1 - No Pain | 9 | 9
  Scar Pain: 2-3 - Mild Pain | 20 | 14
  Scar Pain: 4-6 - Moderate Pain | 13 | 23
  Scar Pain: 7-10 - Severe Pain | 9 | 6
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Neuropathic Categorical Max Pain 36 months; Test type: Superiority or Other; p = 0.076, Mantel Haenszel
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Scar Categorical Max Pain 36 months; Test type: Superiority or Other; p = 0.71, Mantel Haenszel

11. Secondary Outcome: Pain by Visit - Categorical
Description: The subject rated the following questions 'has the scar been painful the past few weeks' and 'have you had any neuropathic pain during the past weeks' on the 1-10 scale were 1 = no, not at all and 10 = yes, very much.
  Pain scale was categorised as 1='no pain', 2-3='mild pain', 4-6='moderate pain', 7-10='severe pain'.
Time Frame: Day 10, Weeks 3, 6, 12, 24, Months 12, 24 and 36
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
Participants
  Day 10: Neuropathic pain: 1: No Pain | 43 | 43
  Day 10: Neuropathic pain: 2-3: Mild Pain | 5 | 4
  Day 10: Neuropathic pain: 4-6: Moderate Pain | 2 | 2
  Day 10: Neuropathic pain: 7-10: Severe Pain | 1 | 3
  Day 10: Scar pain: 1: No Pain | 35 | 32
  Day 10: Scar pain: 2-3: Mild Pain | 10 | 10
  Day 10: Scar pain: 4-6: Moderate Pain | 4 | 9
  Day 10: Scar pain: 7-10: Severe Pain | 2 | 1
  Week 3: Neuropathic pain: number analyzed (Participants) | 50 | 52
  Week 3: Neuropathic pain: 1: No Pain | 44 | 36
  Week 3: Neuropathic pain: 2-3: Mild Pain | 2 | 11
  Week 3: Neuropathic pain: 4-6: Moderate Pain | 3 | 4
  Week 3: Neuropathic pain: 7-10: Severe Pain | 1 | 1
  Week 3: Scar pain: number analyzed (Participants) | 50 | 52
  Week 3: Scar pain: 1: No Pain | 33 | 34
  Week 3: Scar pain: 2-3: Mild Pain | 11 | 14
  Week 3: Scar pain: 4-6: Moderate Pain | 4 | 4
  Week 3: Scar pain: 7-10: Severe Pain | 2 | 0
  Week 6: Neuropathic pain: number analyzed (Participants) | 50 | 51
  Week 6: Neuropathic pain: 1: No Pain | 46 | 42
  Week 6: Neuropathic pain: 2-3: Mild Pain | 2 | 5
  Week 6: Neuropathic pain: 4-6: Moderate Pain | 2 | 3
  Week 6: Neuropathic pain: 7-10: Severe Pain | 0 | 1
  Week 6: Scar pain: number analyzed (Participants) | 50 | 51
  Week 6: Scar pain: 1: No Pain | 35 | 32
  Week 6: Scar pain: 2-3: Mild Pain | 10 | 13
  Week 6: Scar pain: 4-6: Moderate Pain | 5 | 5
  Week 6: Scar pain: 7-10: Severe Pain | 0 | 1
  Week 12: Neuropathic pain: number analyzed (Participants) | 47 | 47
  Week 12: Neuropathic pain: 1: No Pain | 44 | 36
  Week 12: Neuropathic pain: 2-3: Mild Pain | 3 | 5
  Week 12: Neuropathic pain: 4-6: Moderate Pain | 0 | 5
  Week 12: Neuropathic pain: 7-10: Severe Pain | 0 | 1
  Week 12: Scar pain: number analyzed (Participants) | 47 | 48
  Week 12: Scar pain: 1: No Pain | 25 | 30
  Week 12: Scar pain: 2-3: Mild Pain | 16 | 9
  Week 12: Scar pain: 4-6: Moderate Pain | 5 | 8
  Week 12: Scar pain: 7-10: Severe Pain | 1 | 1
  Week 24: Neuropathic pain: number analyzed (Participants) | 47 | 46
  Week 24: Neuropathic pain: 1: No Pain | 44 | 41
  Week 24: Neuropathic pain: 2-3: Mild Pain | 1 | 3
  Week 24: Neuropathic pain: 4-6: Moderate Pain | 2 | 0
  Week 24: Neuropathic pain: 7-10: Severe Pain | 0 | 2
  Week 24: Scar pain: number analyzed (Participants) | 47 | 46
  Week 24: Scar pain: 1: No Pain | 33 | 29
  Week 24: Scar pain: 2-3: Mild Pain | 8 | 9
  Week 24: Scar pain: 4-6: Moderate Pain | 6 | 6
  Week 24: Scar pain: 7-10: Severe Pain | 0 | 2
  Month 12: Neuropathic pain: number analyzed (Participants) | 47 | 48
  Month 12: Neuropathic pain: 1: No Pain | 43 | 40
  Month 12: Neuropathic pain: 2-3: Mild Pain | 2 | 1
  Month 12: Neuropathic pain: 4-6: Moderate Pain | 1 | 4
  Month 12: Neuropathic pain: 7-10: Severe Pain | 1 | 3
  Month 12: Scar pain: number analyzed (Participants) | 47 | 47
  Month 12: Scar pain: 1: No Pain | 30 | 31
  Month 12: Scar pain: 2-3: Mild Pain | 11 | 10
  Month 12: Scar pain: 4-6: Moderate Pain | 2 | 3
  Month 12: Scar pain: 7-10: Severe Pain | 4 | 3
  Month 36: Neuropathic pain: number analyzed (Participants) | 45 | 41
  Month 36: Neuropathic pain: 1: No Pain | 43 | 36
  Month 36: Neuropathic pain: 2-3: Mild Pain | 1 | 2
  Month 36: Neuropathic pain: 4-6: Moderate Pain | 1 | 3
  Month 36: Neuropathic pain: 7-10: Severe Pain | 0 | 0
  Month 36: Scar pain: number analyzed (Participants) | 45 | 41
  Month 36: Scar pain: 1: No Pain | 28 | 25
  Month 36: Scar pain: 2-3: Mild Pain | 12 | 10
  Month 36: Scar pain: 4-6: Moderate Pain | 3 | 4
  Month 36: Scar pain: 7-10: Severe Pain | 2 | 2
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Day 10: Neuropathic pain; Test type: Superiority or Other; p = 0.52, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Day 10: Scar pain; Test type: Superiority or Other; p = 0.44, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 3: Neuropathic pain; Test type: Superiority or Other; p = 0.14, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 3: Scar pain; Test type: Superiority or Other; p = 0.59, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 6: Neuropathic pain; Test type: Superiority or Other; p = 0.17, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 6: Scar pain; Test type: Superiority or Other; p = 0.44, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Neuropathic pain; Test type: Superiority or Other; p = 0.0087, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Scar pain; Test type: Superiority or Other; p = 0.84, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Neuropathic pain; Test type: Superiority or Other; p = 0.43, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Scar pain; Test type: Superiority or Other; p = 0.33, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12 Neuropathic pain; Test type: Superiority or Other; p = 0.21, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12 Scar pain; Test type: Superiority or Other; p = 0.82, Cochran-Mantel-Haenszel
Statistical Analysis 13: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36 Neuropathic pain; Test type: Superiority or Other; p = 0.19, Cochran-Mantel-Haenszel
Statistical Analysis 14: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36 Scar pain; Test type: Superiority or Other; p = 0.77, Cochran-Mantel-Haenszel

12. Secondary Outcome: Soft Tissue Thickening/Overgrowth
Description: The investigator rated the implant site in regards to soft tissue thickening/overgrowth at visits 3-10 according to the following scale:
  0. No soft tissue thickening or overgrowth
  1. Slight soft tissue thickening or overgrowth
  2. Moderate soft tissue thickening or overgrowth. Local treatment and extra controls as indicated*
  3. Marked/distinct soft tissue thickening or overgrowth. Revision surgery is indicated.*
     * Should also be reported on the AE page in the CRF
Time Frame: Day 10, Weeks 3, 6, 12, 24, Months 12, 24 and 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
Participants
  Day 10: No soft tissue thickening | 48 | 52
  Day 10: Slight soft tissue thickening or overgrowth | 2 | 0
  Day 10: Moderate soft tissue thickening or overgrowth | 1 | 0
  Day 10: Marked/distinct soft tissue thickening or overgrow | 0 | 0
  Week 3: number analyzed (Participants) | 50 | 52
  Week 3: No soft tissue thickening | 41 | 50
  Week 3: Slight soft tissue thickening or overgrowth | 6 | 2
  Week 3: Moderate soft tissue thickening or overgrowth | 2 | 0
  Week 3: Marked/distinct soft tissue thickening or overgrow | 1 | 0
  Week 6: number analyzed (Participants) | 50 | 51
  Week 6: No soft tissue thickening | 48 | 48
  Week 6: Slight soft tissue thickening or overgrowth | 1 | 3
  Week 6: Moderate soft tissue thickening or overgrowth | 0 | 0
  Week 6: Marked/distinct soft tissue thickening or overgrow | 1 | 0
  Week 12: number analyzed (Participants) | 47 | 50
  Week 12: No soft tissue thickening | 43 | 43
  Week 12: Slight soft tissue thickening or overgrowth | 4 | 7
  Week 12: Moderate soft tissue thickening or overgrowth | 0 | 0
  Week 12: Marked/distinct soft tissue thickening or overgrow | 0 | 0
  Week 24: number analyzed (Participants) | 47 | 46
  Week 24: No soft tissue thickening | 38 | 42
  Week 24: Slight soft tissue thickening or overgrowth | 8 | 4
  Week 24: Moderate soft tissue thickening or overgrowth | 1 | 0
  Week 24: Marked/distinct soft tissue thickening or overgrow | 0 | 0
  Month 12: number analyzed (Participants) | 48 | 48
  Month 12: No soft tissue thickening | 44 | 44
  Month 12: Slight soft tissue thickening or overgrowth | 1 | 4
  Month 12: Moderate soft tissue thickening or overgrowth | 3 | 0
  Month 12: Marked/distinct soft tissue thickening or overgrow | 0 | 0
  Month 24: number analyzed (Participants) | 46 | 46
  Month 24: No soft tissue thickening | 39 | 41
  Month 24: Slight soft tissue thickening or overgrowth | 6 | 4
  Month 24: Moderate soft tissue thickening or overgrowth | 1 | 1
  Month 24: Marked/distinct soft tissue thickening or overgrow | 0 | 0
  Month 36: number analyzed (Participants) | 45 | 41
  Month 36: No soft tissue thickening | 39 | 37
  Month 36: Slight soft tissue thickening or overgrowth | 6 | 2
  Month 36: Moderate soft tissue thickening or overgrowth | 0 | 2
  Month 36: Marked/distinct soft tissue thickening or overgrow | 0 | 0
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Day 10 Soft tissue thickening/overgrowth; Test type: Superiority or Other; p = 0.12, Mantel Haenszel
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 3 Soft tissue thickening/overgrowth; Test type: Superiority or Other; p = 0.016, Mantel Haenszel
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 6 Soft tissue thickening/overgrowth; Test type: Superiority or Other; p = 0.84, Mantel Haenszel
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12 Soft tissue thickening/overgrowth; Test type: Superiority or Other; p = 0.53, Mantel Haenszel
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24 Soft tissue thickening/overgrowth; Test type: Superiority or Other; p = 0.18, Mantel Haenszel
Statistical Analysis 6: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12 Soft tissue thickening/overgrowth; Test type: Superiority or Other; p = 0.63, Mantel Haenszel
Statistical Analysis 7: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 24 Soft tissue thickening/overgrowth; Test type: Superiority or Other; p = 0.81, Mantel Haenszel
Statistical Analysis 8: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36 Soft tissue thickening/overgrowth; Test type: Superiority or Other; p = 1.00, Mantel Haenszel

13. Secondary Outcome: Visible Abutment Length by Visit for Patients With no Change of Abutment
Description: The investigator measured the visible abutment length at each visit. The length of BA400 test abutments initially placed were longer than BA300 control abutments places. A direct comparison between the groups is not relevant.
  In some cases of increased soft tissue thickening or overgrowth, the abutment was exchanged for a longer abutment. The results presented here are only for patients with no change of abutment
Time Frame: Day 10, Weeks 3, 6, 12, 24, Months 12, 24 and 36
Population: The Intent-to-Treat population (ITT) consisted of all randomised patients with at least one follow-up measurement from visit 3 Day 10 through to visit 10 Month 36.
  This analysis is performed on subjects with no change of abutment.
Measure: Mean (Standard Deviation); unit: millimeters visible abutment length
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 48 | 47
millimeters visible abutment length
  Day 10 | 3.30 (1.23) | 4.17 (1.13)
  Week 3: number analyzed (Participants) | 47 | 47
  Week 3 | 3.34 (1.18) | 3.91 (1.04)
  Week 6: number analyzed (Participants) | 47 | 46
  Week 6 | 4.00 (1.30) | 3.85 (1.13)
  Week 12: number analyzed (Participants) | 44 | 45
  Week 12 | 3.73 (1.35) | 3.51 (1.27)
  Week 24: number analyzed (Participants) | 44 | 41
  Week 24 | 4.07 (1.55) | 3.76 (1.26)
  Month 12: number analyzed (Participants) | 45 | 43
  Month 12 | 4.33 (1.52) | 3.72 (1.20)
  Month 24: number analyzed (Participants) | 43 | 41
  Month 24 | 3.90 (1.61) | 3.56 (1.25)
  Month 36: number analyzed (Participants) | 42 | 37
  Month 36 | 3.74 (1.43) | 3.35 (1.38)
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Visible Abutment Length Day 10; Test type: Superiority or Other; p = 0.0009, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Visible Abutment Length Week 3; Test type: Superiority or Other; p = 0.0080, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Visible Abutment Length Week 6; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Visible Abutment Length Week 12; Test type: Superiority or Other; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Visible Abutment Length Week 24; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Visible Abutment Length Month 12; Test type: Superiority or Other; p = 0.017, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Visible Abutment Length Month 24; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Visible Abutment Length Month 36; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Minimally Invasive Surgery and BA400; Change in Visible Test Abutment - Week 3 change from day 10; Test type: Superiority or Other; p = 0.74, Sign test
Statistical Analysis 10: Comparison: Minimally Invasive Surgery and BA400; Change in Visible Test Abutment - Week 6 change from day 10; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 11: Comparison: Minimally Invasive Surgery and BA400; Change in Visible Test Abutment - Week 12 change from day 10; Test type: Superiority or Other; p = 0.041, Sign test
Statistical Analysis 12: Comparison: Minimally Invasive Surgery and BA400; Change in Visible Test Abutment - Week 24 change from day 10; Test type: Superiority or Other; p = 0.0065, Sign test
Statistical Analysis 13: Comparison: Minimally Invasive Surgery and BA400; Change in Visible Test Abutment - Month 12 change from day 10; Test type: Superiority or Other; p = 0.0003, Sign test
Statistical Analysis 14: Comparison: Minimally Invasive Surgery and BA400; Change in Visible Test Abutment - Month 24 change from day 10; Test type: Superiority or Other; p = 0.028, Sign test
Statistical Analysis 15: Comparison: Minimally Invasive Surgery and BA400; Change in Visible Test Abutment - Month 36 change from day 10; Test type: Superiority or Other; p = 0.037, Sign test
Statistical Analysis 16: Comparison: Traditional Surgery and BA300; Change in Visible Control Abutment - Week 3 change from day 10; Test type: Superiority or Other; p = 0.072, Sign test
Statistical Analysis 17: Comparison: Traditional Surgery and BA300; Change in Visible Control Abutment - Week 6 change from day 10; Test type: Superiority or Other; p = 0.034, Sign test
Statistical Analysis 18: Comparison: Traditional Surgery and BA300; Change in Visible Control Abutment - Week 12 change from day 10; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 19: Comparison: Traditional Surgery and BA300; Change in Visible Control Abutment - Week 24 change from day 10; Test type: Superiority or Other; p = 0.010, Sign test
Statistical Analysis 20: Comparison: Traditional Surgery and BA300; Change in Visible Control Abutment - Month 12 change from day 10; Test type: Superiority or Other; p = 0.0086, Sign test
Statistical Analysis 21: Comparison: Traditional Surgery and BA300; Change in Visible Control Abutment - Month 24 change from day 10; Test type: Superiority or Other; p = 0.0021, Sign test
Statistical Analysis 22: Comparison: Traditional Surgery and BA300; Change in Visible Control Abutment - Month 36 change from day 10; Test type: Superiority or Other; p = 0.0005, Sign test

14. Secondary Outcome: The Aesthetic Outcome of Surgery, the 'Patient and Observer Scar Assessment Scale' Consisted of Two Parts - a Patient and an Observer Scale, Week 12, Month 12 and 36.
Description: The patient scale contains six items (pain, itching, color, stiffness, thickness and irregularity) scored 1-10.
  The observer scale contains six items (vascularity, pigmentation, thickness, relief, pliability and surface area) scored 1-10. Besides the 10-step scale, category boxes are available to score nominal parameters (e.g. type of color).
  Both patient and observer should also score the overall opinion of the scar on the 1-10 scale.
  For all above scales 1=normal skin, 10 worst scar imaginable.
  Total score is the sum of the variables pain, itching, color, stiffness, thickness and irregularity (patient) and vascularity, pigmentation, thickness, relief, pliability and surface area (observer). The scale ranges from 6 to 60 (6 normal, 60 worst scar imaginable).
  The "pain not with in the scar" variable ranges from 1 to 10. 1 being no pain at all and 10 being very much pain
Time Frame: Week 12, Months 12 and 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
units on a scale
  Week 12: Vascularity (observer): number analyzed (Participants) | 47 | 48
  Week 12: Vascularity (observer) | 2.11 (1.15) | 2.81 (1.54)
  Month 12: Vascularity (observer): number analyzed (Participants) | 48 | 47
  Month 12: Vascularity (observer) | 1.98 (1.34) | 2.28 (1.48)
  Month 36: Vascularity (observer): number analyzed (Participants) | 45 | 40
  Month 36: Vascularity (observer) | 1.69 (1.33) | 2.13 (1.49)
  Week 12: Pigmentation (observer): number analyzed (Participants) | 47 | 48
  Week 12: Pigmentation (observer) | 1.96 (1.16) | 2.21 (1.27)
  Month 12: Pigmentation (observer): number analyzed (Participants) | 48 | 47
  Month 12: Pigmentation (observer) | 1.69 (1.26) | 1.91 (1.21)
  Month 36: Pigmentation (observer): number analyzed (Participants) | 45 | 40
  Month 36: Pigmentation (observer) | 1.62 (1.01) | 2.03 (1.61)
  Week 12: Thickness (observer): number analyzed (Participants) | 47 | 48
  Week 12: Thickness (observer) | 2.26 (1.71) | 3.25 (1.49)
  Month 12: Thickness (observer): number analyzed (Participants) | 48 | 47
  Month 12: Thickness (observer) | 2.02 (1.52) | 2.72 (1.99)
  Month 36: Thickness (observer): number analyzed (Participants) | 45 | 40
  Month 36: Thickness (observer) | 2.02 (1.31) | 2.63 (1.85)
  Week 12: Relief (observer): number analyzed (Participants) | 47 | 48
  Week 12: Relief (observer) | 2.11 (1.18) | 3.15 (1.56)
  Month 12: Relief (observer): number analyzed (Participants) | 48 | 47
  Month 12: Relief (observer) | 1.96 (1.24) | 2.74 (1.87)
  Month 36: Relief (observer): number analyzed (Participants) | 45 | 40
  Month 36: Relief (observer) | 1.93 (1.18) | 2.80 (1.86)
  Week 12: Pliability (observer): number analyzed (Participants) | 47 | 48
  Week 12: Pliability (observer) | 2.21 (1.10) | 3.23 (1.75)
  Month 12: Pliability (observer): number analyzed (Participants) | 48 | 47
  Month 12: Pliability (observer) | 2.08 (1.22) | 2.66 (1.70)
  Month 36: Pliability (observer): number analyzed (Participants) | 45 | 40
  Month 36: Pliability (observer) | 1.69 (1.06) | 2.58 (1.60)
  Week 12: Surface Area (observer): number analyzed (Participants) | 47 | 48
  Week 12: Surface Area (observer) | 2.04 (1.12) | 3.06 (1.34)
  Month 12: Surface Area (observer): number analyzed (Participants) | 48 | 47
  Month 12: Surface Area (observer) | 1.94 (1.28) | 2.68 (1.70)
  Month 36: Surface Area (observer): number analyzed (Participants) | 44 | 40
  Month 36: Surface Area (observer) | 1.98 (1.11) | 2.68 (1.62)
  Week 12: Total Score (observer): number analyzed (Participants) | 47 | 48
  Week 12: Total Score (observer) | 12.7 (5.8) | 17.7 (7.4)
  Month 12: Total Score (observer): number analyzed (Participants) | 48 | 47
  Month 12: Total Score (observer) | 11.7 (6.9) | 15.0 (9.0)
  Month 36: Total Score (observer): number analyzed (Participants) | 45 | 40
  Month 36: Total Score (observer) | 10.9 (5.6) | 14.8 (8.9)
  Week 12: Overall Opinion (observer): number analyzed (Participants) | 46 | 46
  Week 12: Overall Opinion (observer) | 2.28 (1.24) | 3.02 (1.22)
  Month 12: Overall Opinion (observer): number analyzed (Participants) | 48 | 47
  Month 12: Overall Opinion (observer) | 2.00 (1.29) | 2.60 (1.65)
  Month 36: Overall Opinion (observer): number analyzed (Participants) | 45 | 40
  Month 36: Overall Opinion (observer) | 1.93 (1.05) | 2.43 (1.52)
  Week 12: Painful (patient): number analyzed (Participants) | 47 | 48
  Week 12: Painful (patient) | 2.00 (1.41) | 2.06 (1.63)
  Month 12: Painful (patient): number analyzed (Participants) | 47 | 47
  Month 12: Painful (patient) | 2.04 (2.01) | 2.02 (1.93)
  Month 36: Painful (patient): number analyzed (Participants) | 45 | 41
  Month 36: Painful (patient) | 1.98 (1.88) | 2.05 (1.83)
  Week 12: Itching (patient): number analyzed (Participants) | 47 | 48
  Week 12: Itching (patient) | 2.49 (2.00) | 2.63 (2.07)
  Month 12: Itching (patient): number analyzed (Participants) | 47 | 47
  Month 12: Itching (patient) | 2.43 (1.98) | 2.45 (2.09)
  Month 36: Itching (patient): number analyzed (Participants) | 45 | 41
  Month 36: Itching (patient) | 2.42 (2.24) | 2.39 (2.07)
  Week 12: Color (patient): number analyzed (Participants) | 44 | 47
  Week 12: Color (patient) | 2.32 (1.49) | 2.06 (1.29)
  Month 12: Color (patient): number analyzed (Participants) | 45 | 46
  Month 12: Color (patient) | 1.78 (1.73) | 1.52 (1.24)
  Month 36: Color (patient): number analyzed (Participants) | 45 | 40
  Month 36: Color (patient) | 1.80 (1.96) | 1.58 (1.63)
  Week 12: Stiffness (patient): number analyzed (Participants) | 46 | 47
  Week 12: Stiffness (patient) | 2.30 (1.71) | 2.47 (1.68)
  Month 12: Stiffness (patient): number analyzed (Participants) | 46 | 47
  Month 12: Stiffness (patient) | 1.76 (1.75) | 1.87 (1.57)
  Month 36: Stiffness (patient): number analyzed (Participants) | 45 | 41
  Month 36: Stiffness (patient) | 1.62 (1.61) | 2.05 (1.60)
  Week 12: Thickness (patient): number analyzed (Participants) | 46 | 47
  Week 12: Thickness (patient) | 2.35 (1.89) | 2.60 (1.64)
  Month 12: Thickness (patient): number analyzed (Participants) | 46 | 47
  Month 12: Thickness (patient) | 1.80 (1.85) | 1.89 (1.62)
  Month 36: Thickness (patient): number analyzed (Participants) | 45 | 40
  Month 36: Thickness (patient) | 2.09 (1.96) | 2.13 (1.68)
  Week 12: Irregularity (patient): number analyzed (Participants) | 45 | 48
  Week 12: Irregularity (patient) | 2.89 (2.14) | 3.27 (2.07)
  Month 12: Irregularity (patient): number analyzed (Participants) | 46 | 47
  Month 12: Irregularity (patient) | 1.87 (1.78) | 2.00 (1.68)
  Month 36: Irregularity (patient): number analyzed (Participants) | 44 | 40
  Month 36: Irregularity (patient) | 1.89 (1.90) | 2.35 (1.97)
  Week 12: Total Score (patient): number analyzed (Participants) | 46 | 48
  Week 12: Total Score (patient) | 13.3 (7.6) | 15.1 (6.5)
  Month 12: Total Score (patient): number analyzed (Participants) | 46 | 47
  Month 12: Total Score (patient) | 11.7 (9.5) | 11.9 (8.1)
  Month 36: Total Score (patient): number analyzed (Participants) | 45 | 40
  Month 36: Total Score (patient) | 11.8 (10.1) | 12.6 (8.7)
  Week 12: Overall Opinion (patient): number analyzed (Participants) | 46 | 48
  Week 12: Overall Opinion (patient) | 2.33 (1.69) | 2.81 (2.13)
  Month 12: Overall Opinion (patient): number analyzed (Participants) | 46 | 47
  Month 12: Overall Opinion (patient) | 1.80 (1.31) | 2.15 (1.53)
  Month 36: Overall Opinion (patient): number analyzed (Participants) | 44 | 40
  Month 36: Overall Opinion (patient) | 1.82 (1.65) | 2.23 (1.79)
  Week 12: Pain not within Scar (patient): number analyzed (Participants) | 47 | 47
  Week 12: Pain not within Scar (patient) | 1.00 (0.00) | 1.62 (1.50)
  Month 12: Pain not within Scar (patient): number analyzed (Participants) | 47 | 48
  Month 12: Pain not within Scar (patient) | 1.09 (0.58) | 1.67 (1.92)
  Month 36: Pain not within Scar (patient): number analyzed (Participants) | 45 | 41
  Month 36: Pain not within Scar (patient) | 1.00 (0.00) | 1.27 (1.03)
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Vascularity (observer); Test type: Superiority or Other; p = 0.026, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Vascularity (observer); Test type: Superiority or Other; p = 0.33, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Vascularity (observer); Test type: Superiority or Other; p = 0.094, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Pigmentation (observer); Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Pigmentation (observer); Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Pigmentation (observer); Test type: Superiority or Other; p = 0.48, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Thickness (observer); Test type: Superiority or Other; p = 0.0003, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Thickness (observer); Test type: Superiority or Other; p = 0.062, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Thickness (observer); Test type: Superiority or Other; p = 0.11, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Relief (observer); Test type: Superiority or Other; p = 0.0003, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Relief (observer); Test type: Superiority or Other; p = 0.079, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Relief (observer); Test type: Superiority or Other; p = 0.025, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Pliability (observer); Test type: Superiority or Other; p = 0.0020, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Pliability (observer); Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Pliability (observer); Test type: Superiority or Other; p = 0.0014, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Surface Area (observer); Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Surface Area (observer); Test type: Superiority or Other; p = 0.023, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Surface Area (observer); Test type: Superiority or Other; p = 0.045, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Total Score (observer); Test type: Superiority or Other; p = 0.0005, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Total Score (observer); Test type: Superiority or Other; p = 0.085, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Total Score (observer); Test type: Superiority or Other; p = 0.030, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Overall Opinion (observer); Test type: Superiority or Other; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Overall Opinion (observer); Test type: Superiority or Other; p = 0.076, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Overall Opinion (observer); Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Painful (patient); Test type: Superiority or Other; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Painful (patient); Test type: Superiority or Other; p = 0.97, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Painful (patient); Test type: Superiority or Other; p = 0.82, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Itching (patient); Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney)
Statistical Analysis 29: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Itching (patient); Test type: Superiority or Other; p = 0.84, Wilcoxon (Mann-Whitney)
Statistical Analysis 30: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Itching (patient); Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney)
Statistical Analysis 31: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Color (patient); Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney)
Statistical Analysis 32: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Color (patient); Test type: Superiority or Other; p = 0.98, Wilcoxon (Mann-Whitney)
Statistical Analysis 33: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Color (patient); Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney)
Statistical Analysis 34: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Stiffness (patient); Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney)
Statistical Analysis 35: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Stiffness (patient); Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 36: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Stiffness (patient); Test type: Superiority or Other; p = 0.017, Wilcoxon (Mann-Whitney)
Statistical Analysis 37: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Thickness (patient); Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney)
Statistical Analysis 38: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Thickness (patient); Test type: Superiority or Other; p = 0.33, Wilcoxon (Mann-Whitney)
Statistical Analysis 39: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Thickness (patient); Test type: Superiority or Other; p = 0.65, Wilcoxon (Mann-Whitney)
Statistical Analysis 40: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Irregularity (patient); Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)
Statistical Analysis 41: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Irregularity (patient); Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 42: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Irregularity (patient); Test type: Superiority or Other; p = 0.080, Wilcoxon (Mann-Whitney)
Statistical Analysis 43: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Total Score (patient); Test type: Superiority or Other; p = 0.28, Wilcoxon (Mann-Whitney)
Statistical Analysis 44: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Total Score (patient); Test type: Superiority or Other; p = 0.44, Wilcoxon (Mann-Whitney)
Statistical Analysis 45: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Total Score (patient); Test type: Superiority or Other; p = 0.19, Wilcoxon (Mann-Whitney)
Statistical Analysis 46: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Overall Opinion (patient); Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney)
Statistical Analysis 47: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Overall Opinion (patient); Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)
Statistical Analysis 48: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Overall Opinion (patient); Test type: Superiority or Other; p = 0.079, Wilcoxon (Mann-Whitney)
Statistical Analysis 49: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Pain not within Scar (patient); Test type: Superiority or Other; p = 0.0018, Wilcoxon (Mann-Whitney)
Statistical Analysis 50: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Pain not within Scar (patient); Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney)
Statistical Analysis 51: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Pain not within Scar (patient); Test type: Superiority or Other; p = 0.068, Wilcoxon (Mann-Whitney)

15. Other Pre Specified Outcome: Health Utilies Index (HUI-III & HUI-II)
Description: Health Utilities Index (HUI) is a generic preference-based system for measuring comprehensive health status and health-related quality of life. Each index provides descriptive evidence on multiple dimensions of life quality.
  HUI3: Comprehensive Health State, Vision, Hearing, Speech, Ambulation, Emotion, Cognition, Pain.
  HUI2: Comprehensive Health State, Sensation, Mobility, Emotion, Cognition, Self Care, Pain.
  Subjects completed HUI2/3 questionnaires at visit 1 (baseline), 7 (week 24), 8 (month 12) and 10 (month 36).
  HUI score of 1 (maximum) describes a state of perfect health. HUI score of 0 describes a state of dead. A negative score of Comprehensive Health State describes a state worse than dead.
Time Frame: baseline (pre-surgery), week 24, months 12 and 36
Population: The Intent-to-Treat population (ITT) consisted of all randomised patients with at least one follow-up measurement from visit 3 Day 10 through to visit 10 month 36.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
units on a scale
  Baseline: Comprehensive Health State (HUI3): number analyzed (Participants) | 45 | 44
  Baseline: Comprehensive Health State (HUI3) | 0.617 (0.272) | 0.620 (0.262)
  Week 24: Comprehensive Health State (HUI3): number analyzed (Participants) | 41 | 41
  Week 24: Comprehensive Health State (HUI3) | 0.705 (0.173) | 0.671 (0.196)
  Month 12: Comprehensive Health State (HUI3): number analyzed (Participants) | 48 | 47
  Month 12: Comprehensive Health State (HUI3) | 0.688 (0.206) | 0.650 (0.232)
  Month 36: Comprehensive Health State (HUI3): number analyzed (Participants) | 43 | 38
  Month 36: Comprehensive Health State (HUI3) | 0.758 (0.147) | 0.639 (0.239)
  Baseline: Vision (HUI3): number analyzed (Participants) | 49 | 51
  Baseline: Vision (HUI3) | 0.952 (0.086) | 0.964 (0.023)
  Week 24: Vision (HUI3): number analyzed (Participants) | 44 | 43
  Week 24: Vision (HUI3) | 0.927 (0.169) | 0.935 (0.126)
  Month 12: Vision (HUI3): number analyzed (Participants) | 48 | 47
  Month 12: Vision (HUI3) | 0.950 (0.087) | 0.940 (0.101)
  Month 36: Vision (HUI3): number analyzed (Participants) | 45 | 39
  Month 36: Vision (HUI3) | 0.942 (0.095) | 0.929 (0.115)
  Baseline: Hearing (HUI3): number analyzed (Participants) | 49 | 47
  Baseline: Hearing (HUI3) | 0.627 (0.304) | 0.601 (0.304)
  Week 24: Hearing (HUI3): number analyzed (Participants) | 45 | 44
  Week 24: Hearing (HUI3) | 0.756 (0.082) | 0.716 (0.089)
  Month 12: Hearing (HUI3): number analyzed (Participants) | 48 | 48
  Month 12: Hearing (HUI3) | 0.726 (0.152) | 0.760 (0.083)
  Month 36: Hearing (HUI3): number analyzed (Participants) | 45 | 41
  Month 36: Hearing (HUI3) | 0.728 (0.172) | 0.683 (0.197)
  Baseline: Speech (HUI3): number analyzed (Participants) | 50 | 50
  Baseline: Speech (HUI3) | 0.913 (0.165) | 0.906 (0.165)
  Week 24: Speech (HUI3): number analyzed (Participants) | 45 | 45
  Week 24: Speech (HUI3) | 0.981 (0.073) | 0.989 (0.055)
  Month 12: Speech (HUI3): number analyzed (Participants) | 48 | 48
  Month 12: Speech (HUI3) | 0.975 (0.078) | 0.975 (0.078)
  Month 36: Speech (HUI3): number analyzed (Participants) | 44 | 40
  Month 36: Speech (HUI3) | 0.984 (0.062) | 0.956 (0.127)
  Baseline: Ambulation (HUI3): number analyzed (Participants) | 50 | 51
  Baseline: Ambulation (HUI3) | 0.983 (0.061) | 0.958 (0.136)
  Week 24: Ambulation (HUI3): number analyzed (Participants) | 45 | 43
  Week 24: Ambulation (HUI3) | 0.989 (0.043) | 0.966 (0.115)
  Month 12: Ambulation (HUI3): number analyzed (Participants) | 48 | 47
  Month 12: Ambulation (HUI3) | 0.990 (0.053) | 0.949 (0.164)
  Month 36: Ambulation (HUI3): number analyzed (Participants) | 45 | 41
  Month 36: Ambulation (HUI3) | 1.000 (0.000) | 0.924 (0.177)
  Baseline: Emotion (HUI3): number analyzed (Participants) | 50 | 51
  Baseline: Emotion (HUI3) | 0.893 (0.170) | 0.945 (0.108)
  Week 24: Emotion (HUI3): number analyzed (Participants) | 45 | 45
  Week 24: Emotion (HUI3) | 0.915 (0.130) | 0.930 (0.090)
  Month 12: Emotion (HUI3): number analyzed (Participants) | 48 | 48
  Month 12: Emotion (HUI3) | 0.911 (0.125) | 0.900 (0.160)
  Month 36: Emotion (HUI3): number analyzed (Participants) | 45 | 41
  Month 36: Emotion (HUI3) | 0.950 (0.073) | 0.906 (0.155)
  Baseline: Cognition (HUI3): number analyzed (Participants) | 47 | 48
  Baseline: Cognition (HUI3) | 0.951 (0.124) | 0.948 (0.144)
  Week 24: Cognition (HUI3): number analyzed (Participants) | 43 | 45
  Week 24: Cognition (HUI3) | 0.966 (0.074) | 0.937 (0.110)
  Month 12: Cognition (HUI3): number analyzed (Participants) | 48 | 47
  Month 12: Cognition (HUI3) | 0.944 (0.133) | 0.909 (0.151)
  Month 36: Cognition (HUI3): number analyzed (Participants) | 44 | 41
  Month 36: Cognition (HUI3) | 0.966 (0.074) | 0.935 (0.108)
  Baseline: Pain (HUI3): number analyzed (Participants) | 50 | 51
  Baseline: Pain (HUI3) | 0.901 (0.174) | 0.918 (0.164)
  Week 24: Pain (HUI3): number analyzed (Participants) | 45 | 46
  Week 24: Pain (HUI3) | 0.933 (0.120) | 0.908 (0.129)
  Month 12: Pain (HUI3): number analyzed (Participants) | 48 | 48
  Month 12: Pain (HUI3) | 0.922 (0.180) | 0.899 (0.215)
  Month 36: Pain (HUI3): number analyzed (Participants) | 45 | 41
  Month 36: Pain (HUI3) | 0.977 (0.054) | 0.926 (0.142)
  Baseline: Comprehensive Health State (HUI2): number analyzed (Participants) | 44 | 44
  Baseline: Comprehensive Health State (HUI2) | 0.799 (0.186) | 0.781 (0.164)
  Week 24: Comprehensive Health State (HUI2): number analyzed (Participants) | 41 | 41
  Week 24: Comprehensive Health State (HUI2) | 0.853 (0.114) | 0.862 (0.099)
  Month 12: Comprehensive Health State (HUI2): number analyzed (Participants) | 48 | 47
  Month 12: Comprehensive Health State (HUI2) | 0.853 (0.114) | 0.827 (0.150)
  Month 36: Comprehensive Health State (HUI2): number analyzed (Participants) | 41 | 38
  Month 36: Comprehensive Health State (HUI2) | 0.896 (0.081) | 0.821 (0.154)
  Baseline: Sensation (HUI2): number analyzed (Participants) | 48 | 47
  Baseline: Sensation (HUI2) | 0.687 (0.264) | 0.666 (0.281)
  Week 24: Sensation (HUI2): number analyzed (Participants) | 44 | 41
  Week 24: Sensation (HUI2) | 0.835 (0.141) | 0.849 (0.066)
  Month 12: Sensation (HUI2): number analyzed (Participants) | 48 | 47
  Month 12: Sensation (HUI2) | 0.822 (0.146) | 0.845 (0.078)
  Month 36: Sensation (HUI2): number analyzed (Participants) | 44 | 39
  Month 36: Sensation (HUI2) | 0.828 (0.148) | 0.809 (0.165)
  Baseline: Mobility (HUI2): number analyzed (Participants) | 50 | 51
  Baseline: Mobility (HUI2) | 0.987 (0.058) | 0.972 (0.093)
  Week 24: Mobility (HUI2): number analyzed (Participants) | 44 | 43
  Week 24: Mobility (HUI2) | 0.995 (0.020) | 0.976 (0.084)
  Month 12: Mobility (HUI2): number analyzed (Participants) | 48 | 47
  Month 12: Mobility (HUI2) | 0.990 (0.057) | 0.965 (0.110)
  Month 36: Mobility (HUI2): number analyzed (Participants) | 45 | 40
  Month 36: Mobility (HUI2) | 1.000 (0.000) | 0.961 (0.105)
  Baseline: Emotion (HUI2): number analyzed (Participants) | 46 | 49
  Baseline: Emotion (HUI2) | 0.912 (0.162) | 0.929 (0.158)
  Week 24: Emotion (HUI2): number analyzed (Participants) | 45 | 46
  Week 24: Emotion (HUI2) | 0.916 (0.138) | 0.940 (0.098)
  Month 12: Emotion (HUI2): number analyzed (Participants) | 48 | 48
  Month 12: Emotion (HUI2) | 0.918 (0.126) | 0.901 (0.140)
  Month 36: Emotion (HUI2): number analyzed (Participants) | 44 | 41
  Month 36: Emotion (HUI2) | 0.959 (0.065) | 0.923 (0.113)
  Baseline: Cognition (HUI2): number analyzed (Participants) | 47 | 48
  Baseline: Cognition (HUI2) | 0.966 (0.072) | 0.960 (0.084)
  Week 24: Cognition (HUI2): number analyzed (Participants) | 43 | 45
  Week 24: Cognition (HUI2) | 0.967 (0.060) | 0.956 (0.066)
  Month 12: Cognition (HUI2): number analyzed (Participants) | 48 | 47
  Month 12: Cognition (HUI2) | 0.971 (0.057) | 0.948 (0.078)
  Month 36: Cognition (HUI2): number analyzed (Participants) | 44 | 41
  Month 36: Cognition (HUI2) | 0.968 (0.059) | 0.092 (0.067)
  Baseline: Self Care (HUI2): number analyzed (Participants) | 47 | 49
  Baseline: Self Care (HUI2) | 0.997 (0.022) | 0.994 (0.030)
  Week 24: Self Care (HUI2): number analyzed (Participants) | 45 | 45
  Week 24: Self Care (HUI2) | 0.997 (0.022) | 0.997 (0.022)
  Month 12: Self Care (HUI2): number analyzed (Participants) | 48 | 47
  Month 12: Self Care (HUI2) | 0.997 (0.022) | 0.987 (0.069)
  Month 36: Self Care (HUI2): number analyzed (Participants) | 45 | 41
  Month 36: Self Care (HUI2) | 1.000 (0.000) | 0.993 (0.033)
  Baseline: Pain (HUI2): number analyzed (Participants) | 49 | 49
  Baseline: Pain (HUI2) | 0.913 (0.224) | 0.956 (0.099)
  Week 24: Pain (HUI2): number analyzed (Participants) | 44 | 45
  Week 24: Pain (HUI2) | 0.957 (0.105) | 0.962 (0.071)
  Month 12: Pain (HUI2): number analyzed (Participants) | 48 | 48
  Month 12: Pain (HUI2) | 0.960 (0.082) | 0.941 (0.146)
  Month 36: Pain (HUI2): number analyzed (Participants) | 44 | 41
  Month 36: Pain (HUI2) | 0.990 (0.020) | 0.924 (0.185)
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Comprehensive Health State (HUI3); Test type: Superiority or Other; p = 0.90, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Comprehensive Health State (HUI3); Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Comprehensive Health State (HUI3); Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Comprehensive Health State (HUI3); Test type: Superiority or Other; p = 0.019, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Vision (HUI3); Test type: Superiority or Other; p = 0.079, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Vision (HUI3); Test type: Superiority or Other; p = 0.96, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Vision (HUI3); Test type: Superiority or Other; p = 0.55, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Vision (HUI3); Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Hearing (HUI3); Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Hearing (HUI3); Test type: Superiority or Other; p = 0.059, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Hearing (HUI3); Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Hearing (HUI3); Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Speech (HUI3); Test type: Superiority or Other; p = 0.73, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Speech (HUI3); Test type: Superiority or Other; p = 0.65, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Speech (HUI3); Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Speech (HUI3); Test type: Superiority or Other; p = 0.35, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Ambulation (HUI3); Test type: Superiority or Other; p = 0.50, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Ambulation (HUI3); Test type: Superiority or Other; p = 0.40, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Ambulation (HUI3); Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Ambulation (HUI3); Test type: Superiority or Other; p = 0.0010, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Emotion (HUI3); Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Emotion (HUI3); Test type: Superiority or Other; p = 0.96, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Emotion (HUI3); Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Emotion (HUI3); Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Cognition (HUI3); Test type: Superiority or Other; p = 0.95, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Cognition (HUI3); Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Cognition (HUI3); Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Cognition (HUI3); Test type: Superiority or Other; p = 0.19, Wilcoxon (Mann-Whitney)
Statistical Analysis 29: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Pain (HUI3); Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney)
Statistical Analysis 30: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Pain (HUI3); Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney)
Statistical Analysis 31: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Pain (HUI3); Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney)
Statistical Analysis 32: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Pain (HUI3); Test type: Superiority or Other; p = 0.040, Wilcoxon (Mann-Whitney)
Statistical Analysis 33: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Comprehensive Health State (HUI2); Test type: Superiority or Other; p = 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 34: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Comprehensive Health State (HUI2); Test type: Superiority or Other; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 35: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Comprehensive Health State (HUI2); Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)
Statistical Analysis 36: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Comprehensive Health State (HUI2); Test type: Superiority or Other; p = 0.0084, Wilcoxon (Mann-Whitney)
Statistical Analysis 37: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Sensation (HUI2); Test type: Superiority or Other; p = 0.77, Wilcoxon (Mann-Whitney)
Statistical Analysis 38: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Sensation (HUI2); Test type: Superiority or Other; p = 0.95, Wilcoxon (Mann-Whitney)
Statistical Analysis 39: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Sensation (HUI2); Test type: Superiority or Other; p = 0.60, Wilcoxon (Mann-Whitney)
Statistical Analysis 40: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Sensation (HUI2); Test type: Superiority or Other; p = 0.48, Wilcoxon (Mann-Whitney)
Statistical Analysis 41: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Mobility (HUI2); Test type: Superiority or Other; p = 0.51, Wilcoxon (Mann-Whitney)
Statistical Analysis 42: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Mobility (HUI2); Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney)
Statistical Analysis 43: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Mobility (HUI2); Test type: Superiority or Other; p = 0.22, Wilcoxon (Mann-Whitney)
Statistical Analysis 44: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Mobility (HUI2); Test type: Superiority or Other; p = 0.0018, Wilcoxon (Mann-Whitney)
Statistical Analysis 45: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Emotion (HUI2); Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney)
Statistical Analysis 46: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Emotion (HUI2); Test type: Superiority or Other; p = 0.52, Wilcoxon (Mann-Whitney)
Statistical Analysis 47: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Emotion (HUI2); Test type: Superiority or Other; p = 0.47, Wilcoxon (Mann-Whitney)
Statistical Analysis 48: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Emotion (HUI2); Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)
Statistical Analysis 49: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Cognition (HUI2); Test type: Superiority or Other; p = 0.82, Wilcoxon (Mann-Whitney)
Statistical Analysis 50: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Cognition (HUI2); Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney)
Statistical Analysis 51: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Cognition (HUI2); Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 52: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Cognition (HUI2); Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 53: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Self Care (HUI2); Test type: Superiority or Other; p = 0.59, Wilcoxon (Mann-Whitney)
Statistical Analysis 54: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Self Care (HUI2); Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney)
Statistical Analysis 55: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Self Care (HUI2); Test type: Superiority or Other; p = 0.55, Wilcoxon (Mann-Whitney)
Statistical Analysis 56: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Self Care (HUI2); Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 57: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Pain (HUI2); Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney)
Statistical Analysis 58: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Pain (HUI2); Test type: Superiority or Other; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 59: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Pain (HUI2); Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)
Statistical Analysis 60: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Pain (HUI2); Test type: Superiority or Other; p = 0.019, Wilcoxon (Mann-Whitney)

16. Other Pre Specified Outcome: Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: The Abbreviated Profile of Hearing Aid Benefit (APHAB) is a 24-item self-assessment, disability-based inventory that can be used to document the outcome of a hearing aid fitting, to compare several fittings, or to evaluate the same fitting over time. The subjects will complete the APHAB at pre-surgery, week 24, month 12 and 36.
  Questions assess 'Ease of Communication', 'Background Noise', 'Reverberation', 'Aversiveness', and 'Global' in the aided and unaided situations. The aided situation was compared to the unaided situation at baseline (pre-surgery).
  For each subscale, a score of 99 indicates that there is 'always' difficulty, and a score of 1 indicated that there is 'never' difficulty for that particular subscale.
Time Frame: Pre-surgery (baseline) to 24 weeks, 12 and 36 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
units on a scale
  Baseline: Ease of Communication (Aided): number analyzed (Participants) | 21 | 26
  Baseline: Ease of Communication (Aided) | 33.9 (22.6) | 21.1 (17.8)
  Baseline: Background Noise (Aided): number analyzed (Participants) | 21 | 26
  Baseline: Background Noise (Aided) | 42.5 (16.3) | 35.5 (23.3)
  Baseline: Reverberation (Aided): number analyzed (Participants) | 19 | 25
  Baseline: Reverberation (Aided) | 48.9 (15.9) | 33.9 (20.3)
  Baseline: Aversiveness (Aided): number analyzed (Participants) | 20 | 25
  Baseline: Aversiveness (Aided) | 35.5 (20.0) | 46.4 (22.8)
  Baseline: Global (Aided): number analyzed (Participants) | 21 | 26
  Baseline: Global (Aided) | 40.8 (17.0) | 30.2 (17.8)
  Baseline: Ease of Communication (Unaided): number analyzed (Participants) | 49 | 48
  Baseline: Ease of Communication (Unaided) | 45.5 (30.4) | 55.4 (26.8)
  Baseline: Background Noise (Unaided): number analyzed (Participants) | 49 | 48
  Baseline: Background Noise (Unaided) | 66.6 (18.4) | 67.4 (19.1)
  Baseline: Reverberation (Unaided): number analyzed (Participants) | 49 | 48
  Baseline: Reverberation (Unaided) | 58.6 (24.7) | 63.0 (25.4)
  Baseline: Aversiveness (Unaided): number analyzed (Participants) | 48 | 48
  Baseline: Aversiveness (Unaided) | 32.2 (24.6) | 25.7 (19.5)
  Baseline: Global (Unaided): number analyzed (Participants) | 49 | 48
  Baseline: Global (Unaided) | 56.9 (20.9) | 61.9 (20.2)
  Baseline: Ease of Communication (Benefit): number analyzed (Participants) | 20 | 23
  Baseline: Ease of Communication (Benefit) | 22.1 (31.5) | 39.9 (26.2)
  Baseline: Background Noise (Benefit): number analyzed (Participants) | 20 | 23
  Baseline: Background Noise (Benefit) | 29.9 (24.3) | 42.0 (26.5)
  Baseline: Reverberation (Benefit): number analyzed (Participants) | 18 | 22
  Baseline: Reverberation (Benefit) | 22.7 (20.6) | 35.9 (29.4)
  Baseline: Aversiveness (Benefit): number analyzed (Participants) | 18 | 22
  Baseline: Aversiveness (Benefit) | -12.3 (24.9) | -23.7 (24.1)
  Baseline: Global (Benefit): number analyzed (Participants) | 20 | 23
  Baseline: Global (Benefit) | 25.3 (20.6) | 39.2 (21.5)
  Week 24: Ease of Communication (Aided): number analyzed (Participants) | 44 | 45
  Week 24: Ease of Communication (Aided) | 20.1 (21.0) | 25.7 (24.8)
  Week 24: Background Noise (Aided): number analyzed (Participants) | 44 | 45
  Week 24: Background Noise (Aided) | 30.5 (13.7) | 33.0 (20.7)
  Week 24: Reverberation (Aided): number analyzed (Participants) | 44 | 44
  Week 24: Reverberation (Aided) | 29.4 (12.4) | 34.9 (19.8)
  Week 24: Aversiveness (Aided): number analyzed (Participants) | 44 | 45
  Week 24: Aversiveness (Aided) | 42.9 (21.9) | 44.7 (26.2)
  Week 24: Global (Aided): number analyzed (Participants) | 44 | 45
  Week 24: Global (Aided) | 26.7 (13.0) | 31.1 (18.8)
  Week 24: Ease of Communication (Unaided): number analyzed (Participants) | 28 | 25
  Week 24: Ease of Communication (Unaided) | 44.2 (26.6) | 52.8 (28.8)
  Week 24: Background Noise (Unaided): number analyzed (Participants) | 28 | 25
  Week 24: Background Noise (Unaided) | 66.5 (17.8) | 65.3 (19.3)
  Week 24: Reverberation (Unaided): number analyzed (Participants) | 28 | 25
  Week 24: Reverberation (Unaided) | 57.1 (21.4) | 63.2 (19.6)
  Week 24: Aversiveness (Unaided): number analyzed (Participants) | 28 | 25
  Week 24: Aversiveness (Unaided) | 29.6 (22.3) | 18.3 (17.5)
  Week 24: Global (Unaided): number analyzed (Participants) | 28 | 25
  Week 24: Global (Unaided) | 55.9 (18.6) | 60.4 (19.3)
  Week 24: Ease of Communication (Benefit): number analyzed (Participants) | 43 | 41
  Week 24: Ease of Communication (Benefit) | 29.3 (30.6) | 30.6 (36.5)
  Week 24: Background Noise (Benefit): number analyzed (Participants) | 43 | 41
  Week 24: Background Noise (Benefit) | 37.8 (22.8) | 37.6 (22.8)
  Week 24: Reverberation (Benefit): number analyzed (Participants) | 43 | 41
  Week 24: Reverberation (Benefit) | 31.5 (24.1) | 32.4 (32.7)
  Week 24: Aversiveness (Benefit): number analyzed (Participants) | 42 | 41
  Week 24: Aversiveness (Benefit) | -10.7 (31.2) | -20.4 (25.3)
  Week 24: Global (Benefit): number analyzed (Participants) | 43 | 41
  Week 24: Global (Benefit) | 32.9 (21.0) | 33.5 (26.5)
  Month 12: Ease of Communication (Aided): number analyzed (Participants) | 47 | 47
  Month 12: Ease of Communication (Aided) | 17.5 (18.0) | 19.7 (18.7)
  Month 12: Background Noise (Aided): number analyzed (Participants) | 48 | 47
  Month 12: Background Noise (Aided) | 29.9 (14.8) | 32.3 (14.1)
  Month 12: Reverberation (Aided): number analyzed (Participants) | 48 | 47
  Month 12: Reverberation (Aided) | 31.8 (16.5) | 30.9 (14.0)
  Month 12: Aversiveness (Aided): number analyzed (Participants) | 47 | 47
  Month 12: Aversiveness (Aided) | 39.3 (23.0) | 37.4 (28.8)
  Month 12: Global (Aided): number analyzed (Participants) | 48 | 47
  Month 12: Global (Aided) | 26.7 (13.5) | 27.6 (12.2)
  Month 12: Ease of Communication (Unaided): number analyzed (Participants) | 27 | 28
  Month 12: Ease of Communication (Unaided) | 41.8 (27.5) | 52.0 (28.5)
  Month12: Background Noise (Unaided): number analyzed (Participants) | 27 | 29
  Month12: Background Noise (Unaided) | 65.0 (20.8) | 64.1 (19.7)
  Month 12: Reverberation (Unaided): number analyzed (Participants) | 28 | 28
  Month 12: Reverberation (Unaided) | 53.4 (20.0) | 60.9 (20.0)
  Month12: Aversiveness (Unaided): number analyzed (Participants) | 27 | 29
  Month12: Aversiveness (Unaided) | 30.2 (21.8) | 23.5 (20.7)
  Month 12: Global (Unaided): number analyzed (Participants) | 28 | 29
  Month 12: Global (Unaided) | 53.7 (20.4) | 58.7 (19.9)
  Month 12: Ease of Communication (Benefit): number analyzed (Participants) | 27 | 28
  Month 12: Ease of Communication (Benefit) | 41.8 (27.5) | 52.0 (28.5)
  Month 12: Background Noise (Benefit): number analyzed (Participants) | 27 | 29
  Month 12: Background Noise (Benefit) | 65.0 (20.8) | 64.1 (19.7)
  Month 12: Reverberation (Benefit): number analyzed (Participants) | 28 | 28
  Month 12: Reverberation (Benefit) | 53.4 (20.0) | 60.9 (20.0)
  Month 12: Aversiveness (Benefit): number analyzed (Participants) | 27 | 29
  Month 12: Aversiveness (Benefit) | 30.2 (21.8) | 23.5 (20.7)
  Month 12: Global (Benefit): number analyzed (Participants) | 28 | 29
  Month 12: Global (Benefit) | 53.7 (20.4) | 58.7 (19.9)
  Month 36: Ease of Communication (Aided): number analyzed (Participants) | 45 | 41
  Month 36: Ease of Communication (Aided) | 19.3 (21.3) | 18.1 (20.1)
  Month 36: Background Noise (Aided): number analyzed (Participants) | 45 | 41
  Month 36: Background Noise (Aided) | 33.5 (16.6) | 35.7 (17.2)
  Month 36: Reverberation (Aided): number analyzed (Participants) | 45 | 41
  Month 36: Reverberation (Aided) | 32.7 (18.2) | 30.6 (13.9)
  Month 36: Aversiveness (Aided): number analyzed (Participants) | 45 | 41
  Month 36: Aversiveness (Aided) | 36.2 (24.8) | 36.9 (25.9)
  Month 36: Global (Aided): number analyzed (Participants) | 45 | 41
  Month 36: Global (Aided) | 28.5 (15.8) | 28.1 (14.2)
  Month 36: Ease of Communication (Unaided): number analyzed (Participants) | 26 | 26
  Month 36: Ease of Communication (Unaided) | 45.9 (23.6) | 50.0 (23.8)
  Month 36: Background Noise (Unaided): number analyzed (Participants) | 27 | 26
  Month 36: Background Noise (Unaided) | 66.5 (19.4) | 62.9 (18.3)
  Month 36: Reverberation (Unaided): number analyzed (Participants) | 27 | 26
  Month 36: Reverberation (Unaided) | 60.4 (21.1) | 56.6 (19.6)
  Month 36: Aversiveness (Unaided): number analyzed (Participants) | 26 | 26
  Month 36: Aversiveness (Unaided) | 38.5 (23.0) | 26.1 (20.8)
  Month 36: Global (Unaided): number analyzed (Participants) | 27 | 26
  Month 36: Global (Unaided) | 57.7 (18.1) | 56.5 (17.3)
  Month 36: Ease of Communication (Benefit): number analyzed (Participants) | 44 | 38
  Month 36: Ease of Communication (Benefit) | 27.6 (36.6) | 38.5 (28.0)
  Month 36: Background Noise (Benefit): number analyzed (Participants) | 44 | 38
  Month 36: Background Noise (Benefit) | 32.8 (21.1) | 33.9 (22.2)
  Month 36: Reverberation (Benefit): number analyzed (Participants) | 44 | 38
  Month 36: Reverberation (Benefit) | 27.8 (26.8) | 34.2 (30.6)
  Month 36: Aversiveness (Benefit): number analyzed (Participants) | 43 | 38
  Month 36: Aversiveness (Benefit) | -2.22 (31.71) | -9.19 (32.95)
  Month 36: Global (Benefit): number analyzed (Participants) | 44 | 38
  Month 36: Global (Benefit) | 29.4 (23.1) | 35.5 (22.8)
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Ease of Communication (Aided); Test type: Superiority or Other; p = 0.047, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Background Noise (Aided); Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Reverberation (Aided); Test type: Superiority or Other; p = 0.015, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Aversiveness (Aided); Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Global (Aided); Test type: Superiority or Other; p = 0.041, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Ease of Communication (Unaided); Test type: Superiority or Other; p = 0.071, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Background Noise (Unaided); Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Reverberation (Unaided); Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Aversiveness (Unaided); Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Global (Unaided); Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Ease of Communication (Benefit); Test type: Superiority or Other; p = 0.12, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Background Noise (Benefit); Test type: Superiority or Other; p = 0.19, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Reverberation (Benefit); Test type: Superiority or Other; p = 0.055, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Aversiveness (Benefit); Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Global (Benefit); Test type: Superiority or Other; p = 0.042, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Ease of Communication (Aided); Test type: Superiority or Other; p = 0.19, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Background Noise (Aided); Test type: Superiority or Other; p = 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Reverberation (Aided); Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Aversiveness (Aided); Test type: Superiority or Other; p = 0.73, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Global (Aided); Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Ease of Communication (Unaided); Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Background Noise (Unaided); Test type: Superiority or Other; p = 0.81, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Reverberation (Unaided); Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Aversiveness (Unaided); Test type: Superiority or Other; p = 0.038, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Global (Unaided); Test type: Superiority or Other; p = 0.53, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Ease of Communication (Benefit); Test type: Superiority or Other; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Background Noise (Benefit); Test type: Superiority or Other; p = 0.83, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Reverberation (Benefit); Test type: Superiority or Other; p = 0.71, Wilcoxon (Mann-Whitney)
Statistical Analysis 29: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Aversiveness (Benefit); Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney)
Statistical Analysis 30: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 24: Global (Benefit); Test type: Superiority or Other; p = 0.81, Wilcoxon (Mann-Whitney)
Statistical Analysis 31: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Ease of Communication (Aided); Test type: Superiority or Other; p = 0.51, Wilcoxon (Mann-Whitney)
Statistical Analysis 32: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Background Noise (Aided); Test type: Superiority or Other; p = 0.47, Wilcoxon (Mann-Whitney)
Statistical Analysis 33: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Reverberation (Aided); Test type: Superiority or Other; p = 0.93, Wilcoxon (Mann-Whitney)
Statistical Analysis 34: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Aversiveness (Aided); Test type: Superiority or Other; p = 0.62, Wilcoxon (Mann-Whitney)
Statistical Analysis 35: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Global (Aided); Test type: Superiority or Other; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 36: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Ease of Communication (Unaided); Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)
Statistical Analysis 37: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Background Noise (Unaided); Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney)
Statistical Analysis 38: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Reverberation (Unaided); Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney)
Statistical Analysis 39: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Aversiveness (Unaided); Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney)
Statistical Analysis 40: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Global (Unaided); Test type: Superiority or Other; p = 0.40, Wilcoxon (Mann-Whitney)
Statistical Analysis 41: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Ease of Communication (Benefit); Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney)
Statistical Analysis 42: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Background Noise (Benefit); Test type: Superiority or Other; p = 0.90, Wilcoxon (Mann-Whitney)
Statistical Analysis 43: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Reverberation (Benefit); Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 44: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Aversiveness (Benefit); Test type: Superiority or Other; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 45: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Global (Benefit); Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney)
Statistical Analysis 46: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Ease of Communication (Aided); Test type: Superiority or Other; p = 0.84, Wilcoxon (Mann-Whitney)
Statistical Analysis 47: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Background Noise (Aided); Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)
Statistical Analysis 48: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Reverberation (Aided); Test type: Superiority or Other; p = 0.71, Wilcoxon (Mann-Whitney)
Statistical Analysis 49: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Aversiveness (Aided); Test type: Superiority or Other; p = 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 50: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Global (Aided); Test type: Superiority or Other; p = 0.78, Wilcoxon (Mann-Whitney)
Statistical Analysis 51: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Ease of Communication (Unaided); Test type: Superiority or Other; p = 0.50, Wilcoxon (Mann-Whitney)
Statistical Analysis 52: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Background Noise (Unaided); Test type: Superiority or Other; p = 0.48, Wilcoxon (Mann-Whitney)
Statistical Analysis 53: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Reverberation (Unaided); Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)
Statistical Analysis 54: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Aversiveness (Unaided); Test type: Superiority or Other; p = 0.041, Wilcoxon (Mann-Whitney)
Statistical Analysis 55: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Global (Unaided); Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney)
Statistical Analysis 56: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Ease of Communication (Benefit); Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 57: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Background Noise (Benefit); Test type: Superiority or Other; p = 0.48, Wilcoxon (Mann-Whitney)
Statistical Analysis 58: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Reverberation (Benefit); Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)
Statistical Analysis 59: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Aversiveness (Benefit); Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)
Statistical Analysis 60: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Global (Benefit); Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney)

17. Other Pre Specified Outcome: Use of Sound Processor
Description: Use of the sound processor can be seen as a reflection of patient satisfaction and treatment compliance. Patients were asked to record how many hours per week they used the sound processor after Baha loading at week 3.
Time Frame: Weeks 6, 12, 24, Months 12, 24, 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours of use per week
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
Hours of use per week
  Week 6: No Sound Processor Usage (Patients): number analyzed (Participants) | 50 | 51
  Week 6: No Sound Processor Usage (Patients) | 0 (0) | 0 (0)
  Week 6: Sound Processor Usage (hours/week): number analyzed (Participants) | 50 | 51
  Week 6: Sound Processor Usage (hours/week) | 80.4 (30.1) | 83.6 (27.7)
  Week 12: No Sound Processor Usage (Patients): number analyzed (Participants) | 47 | 50
  Week 12: No Sound Processor Usage (Patients) | 2 (4.8) | 1 (2.1)
  Week 12: Sound Processor Usage (hours/week): number analyzed (Participants) | 47 | 50
  Week 12: Sound Processor Usage (hours/week) | 75.2 (33.0) | 77.9 (29.7)
  Week 24: No Sound Processor Usage (Patients): number analyzed (Participants) | 47 | 46
  Week 24: No Sound Processor Usage (Patients) | 1 (2.1) | 0 (0)
  Week 24: Sound Processor Usage (hours/week): number analyzed (Participants) | 47 | 46
  Week 24: Sound Processor Usage (hours/week) | 74.6 (34.1) | 78.0 (30.6)
  Month 12: No Sound Processor Usage (Patients): number analyzed (Participants) | 48 | 48
  Month 12: No Sound Processor Usage (Patients) | 2 (4.2) | 1 (2.1)
  Month 12: Sound Processor Usage (hours/week): number analyzed (Participants) | 48 | 48
  Month 12: Sound Processor Usage (hours/week) | 73.5 (35.1) | 80.1 (29.4)
  Month 24: No Sound Processor Usage (Patients): number analyzed (Participants) | 46 | 46
  Month 24: No Sound Processor Usage (Patients) | 2 (4.3) | 1 (2.3)
  Month 24: Sound Processor Usage (hours/week): number analyzed (Participants) | 46 | 46
  Month 24: Sound Processor Usage (hours/week) | 68.3 (36.7) | 72.1 (36.6)
  Month 36: No Sound Processor Usage (Patients): number analyzed (Participants) | 45 | 41
  Month 36: No Sound Processor Usage (Patients) | 0 (0) | 1 (2.4)
  Month 36: Sound Processor Usage (hours/week): number analyzed (Participants) | 45 | 41
  Month 36: Sound Processor Usage (hours/week) | 74.3 (32.2) | 77.7 (32.6)
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Sound Processor Usage: Week 6; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Use of Sound Processor: Week 12; Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Use of Sound Processor: Week 24; Test type: Superiority or Other; p = 0.83, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Use of Sound Processor: Month 12; Test type: Superiority or Other; p = 0.52, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Use of Sound Processor: Month 24; Test type: Superiority or Other; p = 0.67, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Use of Sound Processor: Month 36; Test type: Superiority or Other; p = 0.71, Wilcoxon (Mann-Whitney)

18. Other Pre Specified Outcome: Implant Stability (ISQ)
Description: ISQ is a well-established method to measure stability of osseointegrated implants and has been used for several years both for bone conduction implants and for dental implants. Measurements were performed using resonance frequency analysis at the abutment level. The highest and lowest ISQ value out of two perpendicular measurements obtained at each time point was recorded, ISQ High and ISQ Low. The ISQ values ranges from 1 to 100.
  Overall, the length of test abutments (BA400) were longer than control abutments (BA300) and there is an inverse correlation between abutment length and stability. A direct comparison between the groups is not relevant.
  Implant Stability Quotient (ISQ) was recorded at surgery as a baseline value and at visit 2-10.
Time Frame: Surgery, Day 10, Weeks 3, 6, 12, 24, Months 12, 24, 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Implant Stability Quotient
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
Implant Stability Quotient
  Surgery: ISQ (High) | 55.4 (6.6) | 66.2 (4.1)
  Surgery: ISQ (Low) | 53.2 (6.7) | 64.1 (4.8)
  Day 10: ISQ (High) | 54.9 (8.7) | 63.4 (9.3)
  Day 10: ISQ (Low) | 52.6 (9.8) | 61.3 (9.7)
  Week 3: ISQ (High): number analyzed (Participants) | 50 | 52
  Week 3: ISQ (High) | 54.6 (9.0) | 65.2 (5.2)
  Week 3: ISQ (Low): number analyzed (Participants) | 50 | 52
  Week 3: ISQ (Low) | 52.2 (9.9) | 63.3 (5.8)
  Week 6: ISQ (High): number analyzed (Participants) | 50 | 51
  Week 6: ISQ (High) | 56.6 (7.3) | 64.6 (6.9)
  Week 6: ISQ (Low): number analyzed (Participants) | 50 | 51
  Week 6: ISQ (Low) | 53.3 (9.3) | 62.4 (7.9)
  Week 12: ISQ (High): number analyzed (Participants) | 47 | 50
  Week 12: ISQ (High) | 58.0 (6.3) | 66.1 (4.9)
  Week 12: ISQ (Low): number analyzed (Participants) | 47 | 50
  Week 12: ISQ (Low) | 55.6 (6.7) | 63.8 (6.0)
  Week 24: ISQ (High): number analyzed (Participants) | 47 | 46
  Week 24: ISQ (High) | 59.7 (5.4) | 66.8 (4.3)
  Week 24: ISQ (Low): number analyzed (Participants) | 47 | 46
  Week 24: ISQ (Low) | 57.5 (5.7) | 64.4 (5.3)
  Month 12: ISQ (High): number analyzed (Participants) | 48 | 48
  Month 12: ISQ (High) | 59.6 (5.0) | 67.6 (4.0)
  Month 12: ISQ (Low): number analyzed (Participants) | 48 | 48
  Month 12: ISQ (Low) | 58.0 (4.8) | 65.5 (4.7)
  Month 24: ISQ (High): number analyzed (Participants) | 46 | 46
  Month 24: ISQ (High) | 60.4 (6.1) | 66.8 (5.5)
  Month 24: ISQ (Low): number analyzed (Participants) | 46 | 46
  Month 24: ISQ (Low) | 59.0 (6.2) | 66.2 (4.3)
  Month 36: ISQ (High): number analyzed (Participants) | 45 | 41
  Month 36: ISQ (High) | 59.6 (6.0) | 67.0 (5.3)
  Month 36: ISQ (Low): number analyzed (Participants) | 45 | 41
  Month 36: ISQ (Low) | 58.2 (5.8) | 62.5 (5.5)

19. Other Pre Specified Outcome: Smoking Habits by Visit
Description: Nicotine use and smoking habits were recorded for patients.
  1. Does not smoke
  2. Less than 10 cigarettes/day (Low consumption)
  3. Between 11 and 20 cigarettes/day (Medium consumption)
  4. Between 21 and 40 cigarettes/day (High consumption)
  5. More than 40 cigarettes/day (Very high consumption)
  In Sweden a large proportion of adults use another form of tobacco, wet snuff. In Sweden the patients were asked if they used wet snuff.
Time Frame: baseline, Weeks 3, 12, Months 12, 24 and 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 51 | 52
Participants
  Baseline Smoking: No Smoking | 37 | 38
  Baseline Smoking: Yes, Less than 10 cigarettes/day | 5 | 3
  Baseline Smoking: Yes, Between 11-20 cigarettes/day | 8 | 8
  Baseline Smoking: Yes, Between 21-40 cigarettes/day | 1 | 2
  Baseline Smoking: Yes, More than 40 cigarettes/day | 0 | 0
  Baseline Smoking: Wet Snuff | 0 | 0
  Baseline Smoking: Not answered | 0 | 1
  Week 3 Smoking: number analyzed (Participants) | 50 | 52
  Week 3 Smoking: No Smoking | 36 | 39
  Week 3 Smoking: Yes, Less than 10 cigarettes/day | 5 | 4
  Week 3 Smoking: Yes, Between 11-20 cigarettes/day | 7 | 7
  Week 3 Smoking: Yes, Between 21-40 cigarettes/day | 1 | 1
  Week 3 Smoking: Yes, More than 40 cigarettes/day | 0 | 0
  Week 3 Smoking: Wet Snuff | 1 | 0
  Week 3 Smoking: Not answered | 0 | 1
  Week 12 Smoking: number analyzed (Participants) | 47 | 50
  Week 12 Smoking: No Smoking | 32 | 38
  Week 12 Smoking: Yes, Less than 10 cigarettes/day | 8 | 4
  Week 12 Smoking: Yes, Between 11-20 cigarettes/day | 4 | 6
  Week 12 Smoking: Yes, Between 21-40 cigarettes/day | 2 | 2
  Week 12 Smoking: Yes, More than 40 cigarettes/day | 0 | 0
  Week 12 Smoking: Wet Snuff | 1 | 0
  Week 12 Smoking: Not answered | 0 | 0
  Month 12 Smoking: number analyzed (Participants) | 48 | 48
  Month 12 Smoking: No Smoking | 35 | 33
  Month 12 Smoking: Yes, Less than 10 cigarettes/day | 8 | 4
  Month 12 Smoking: Yes, Between 11-20 cigarettes/day | 2 | 8
  Month 12 Smoking: Yes, Between 21-40 cigarettes/day | 2 | 3
  Month 12 Smoking: Yes, More than 40 cigarettes/day | 0 | 0
  Month 12 Smoking: Wet Snuff | 1 | 0
  Month 12 Smoking: Not answered | 0 | 0
  Month 24 Smoking: number analyzed (Participants) | 46 | 46
  Month 24 Smoking: No Smoking | 34 | 31
  Month 24 Smoking: Yes, Less than 10 cigarettes/day | 7 | 6
  Month 24 Smoking: Yes, Between 11-20 cigarettes/day | 3 | 6
  Month 24 Smoking: Yes, Between 21-40 cigarettes/day | 1 | 3
  Month 24 Smoking: Yes, More than 40 cigarettes/day | 0 | 0
  Month 24 Smoking: Wet Snuff | 0 | 0
  Month 24 Smoking: Not answered | 1 | 0
  Month 36 Smoking: number analyzed (Participants) | 45 | 41
  Month 36 Smoking: No Smoking | 34 | 30
  Month 36 Smoking: Yes, Less than 10 cigarettes/day | 6 | 3
  Month 36 Smoking: Yes, Between 11-20 cigarettes/day | 4 | 6
  Month 36 Smoking: Yes, Between 21-40 cigarettes/day | 1 | 2
  Month 36 Smoking: Yes, More than 40 cigarettes/day | 0 | 0
  Month 36 Smoking: Wet Snuff | 0 | 0
  Month 36 Smoking: Not answered | 0 | 0
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Baseline: Smoking and Wet Snuff habits; Test type: Superiority or Other; p = 0.91, Mantel Haenszel
Statistical Analysis 2: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 3: Smoking and Wet Snuff habits; Test type: Superiority or Other; p = 0.70, Mantel Haenszel
Statistical Analysis 3: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Week 12: Smoking and Wet Snuff habits; Test type: Superiority or Other; p = 0.95, Mantel Haenszel
Statistical Analysis 4: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 12: Smoking and Wet Snuff habits; Test type: Superiority or Other; p = 0.22, Mantel Haenszel
Statistical Analysis 5: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 24: Smoking and Wet Snuff habits; Test type: Superiority or Other; p = 0.19, Mantel Haenszel
Statistical Analysis 6: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Month 36: Smoking and Wet Snuff habits; Test type: Superiority or Other; p = 0.45, Mantel Haenszel

20. Other Pre Specified Outcome: Loss of Implant
Description: 'Loss of Implant' refers to the loss of the implant for reasons including failure of implant to osseointegrate, or an implant that was loose form surgery. It does not include elected removal of the device.
Time Frame: from surgery through to 36 months
Population: The Safety Population includes all patients who had the surgical treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 52 | 52
Participants | 1 | 1
Statistical Analysis 1: Comparison: Minimally Invasive Surgery and BA400 vs Traditional Surgery and BA300; Loss of Implant (safety population); Test type: Superiority or Other; p = 0.989, Log Rank; Hazard Ratio (HR) = 0.98

21. Other Pre Specified Outcome: Removal of Abutment
Description: Count of subjects who had their abutment removed for reasons of health and safety, such as infection, inflammation or pain.
Time Frame: from surgery through to 36 months
Population: The Safety Population includes all patients who had the surgical treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
Number analyzed (Participants) | 52 | 52
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: 3 years
Description: One subject was randomised to control group (BA300) but received the test abutment. The subject was considered as an 'Early withdrawal' after surgery. The Number of Participants at Risk for All-Cause Mortality is therefore greater than the number Started in the Participant Flow, though the subject was still included in the safety population.
Arm/Group | Minimally Invasive Surgery and BA400 | Traditional Surgery and BA300
All-Cause Mortality (participants affected / at risk) | 1/52 | 1/52
Serious Adverse Events (participants affected / at risk) | 7/52 | 10/52
Other Adverse Events (participants affected / at risk) | 35/52 | 39/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minimally Invasive Surgery and BA400 (N=52) | Traditional Surgery and BA300 (N=52)
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 1 (2)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Implant site pain (General disorders) | 0 (0) | 2 (2)
Device Expulsion (General disorders) | 0 (0) | 1 (1)
Accidental Death (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Ear operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Mastoidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Device failure (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minimally Invasive Surgery and BA400 (N=52) | Traditional Surgery and BA300 (N=52)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Implant site pain (Gastrointestinal disorders) | 2 (3) | 5 (6)
Implant site scar (General disorders) | 2 (2) | 4 (4)
Installation site erythema (General disorders) | 25 (57) | 18 (29)
Ear Infection (Infections and infestations) | 1 (1) | 4 (5)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4)
Otitis media (Infections and infestations) | 0 (0) | 4 (4)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 6 (9)
Wound secretions (Injury, poisoning and procedural complications) | 19 (34) | 12 (16)
Dizzy postural (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 3 (4)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 8 (12) | 3 (3)
Excessive skin (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Skin swelling (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
The Holgers Index was developed to assess the soft tissue status in relation to soft tissue reduction surgery, not tissue preservation surgery. There is community discussion as to whether it is appropriate for preservation surgery analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-07-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT01796236/SAP_000.pdf
  • Study Protocol (2013-09-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT01796236/Prot_001.pdf